CLINICAL TRIAL: NCT06996158
Title: Prospective Evaluation Assessing Performance, Survivorship and Patient Reported Outcome Measures of Mobile Bearing Total Knee System (U2 MB™ Knee).
Brief Title: Prospective Evaluation Assessing U2 MB™ Total Knee System
Status: Not yet recruiting | Type: Observational
Sponsor: MSK Doctors & Associates Ltd (Industry)
Collaborators: United Orthopedics Inc. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 25/WM/0048
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis; Musculoskeletal Abnormalities
MeSH Terms: conditions — Osteoarthritis; Musculoskeletal Abnormalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 13 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Knee implant group

SUMMARY:
The goal of this study is to evaluate the safety and effectiveness of the United Orthopaedics Mobile Bearing Total Knee System (U2 MB™ Knee) in patients undergoing total knee replacement surgery due to end-stage knee osteoarthritis. The main questions it aims to answer are:

1. What is the component survivorship of the U2 MB™ Knee system at 1, 3, 5, and 10 years?

Participants will:

1. Return for follow-up assessments at Year 1, Year 3, Year 5, and Year 10 after surgery
2. Undergo clinical evaluations including functional outcome scoring, radiographic imaging.

This study will take place across three investigational sites and will involve 150 knee replacements using U2 MB™ components. The study's objectives include assessing early to long-term outcomes in terms of implant survivorship, clinical function, patient satisfaction, radiological findings, and overall safety of the device over a 10-year period.

DETAILED DESCRIPTION:
Non-interventional prospective follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. All patients suitable for a cemented Total Knee Replacement, MBC design
2. All elective pathology (including Osteoarthritis, Rheumatoid arthritis, Post-traumatic arthritis not requiring stemmed components, Avascular necrosis)
3. Willing to voluntarily sign the informed consent form
4. Willing and able to comply with the protocol, able to read and complete the required forms, and willing and able to adhere to the requirements of the protocol through the 10-year postoperative follow-up visit.

Exclusion Criteria:

1. Skeletally immature (less than 21 years of age) at time of implantation
2. Active native knee joint infection
3. Post-traumatic arthritis requiring stemmed components
4. Malignancy around the knee
5. All patients who are personally unable to take part in fully informed consent (dementia, reduced AMTS etc)
6. Patients who will not be available to return for the predetermined appointments in order to complete the 10 years follow-up
7. Has inadequate neuromuscular status (e.g., prior paralysis, fusion, and/or inadequate abductor strength), poor bone stock, poor skin coverage around the joint which would make the procedure unjustifiable
8. Currently enrolled in another clinical investigation which could affect the endpoints of this protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2038-05-27 (Estimated); Study Completion 2038-11-30 (Estimated)

PRIMARY OUTCOMES:
Study of the survivorship of the U2 MB™ Knee system and its components, defined as no removal or revision of any components during a 10-year interval after implantation. | 10 years

SECONDARY OUTCOMES:
Two standardized scores will grade the functional score of the knee joint over time: Knee Society Score (KSS) and Oxford Knee Score (OKS) | 10 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800